CLINICAL TRIAL: NCT05269706
Title: Cannabidiol in the Treatment of Opioid Use Disorder
Brief Title: Investigation of the Pharmacokinetic Profile of CBD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yasmin Hurd (Other)
Responsible Party: Sponsor-Investigator, Yasmin Hurd, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STUDY-19-00681
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder
Keywords: Methadone; Buprenorphine; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Study will be conducted using a cross-over design, separated by a 1-week washout period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Meal (Experimental): Participants taking a standard meal.
  Interventions: Drug: Cannabidiol 200mg; Drug: Epidiolex; Drug: Cannabidiol 400mg; Drug: Placebo
- High Fat Meal (Experimental): Participants taking a high fat meal.
  Interventions: Drug: Cannabidiol 200mg; Drug: Epidiolex; Drug: Cannabidiol 400mg; Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol 200mg — Cannabidiol 200mg (twice daily)
  Other Names: BSPG CBD
Drug: Epidiolex — Epidiolex 400mg (twice daily)
Drug: Cannabidiol 400mg — Cannabidiol 400mg (twice daily)
  Other Names: BSPG CBD
Drug: Placebo — Matching Placebo (Twice Daily)

SUMMARY:
The goal of the current study is to evaluate the bioavailability of CBD in normal healthy Individuals. This is an open cross-overdesign study in healthy individuals to assess the safety and pharmacokinetic (PK) effects of cannabidiol.

DETAILED DESCRIPTION:
The goal of this study is to determine the pharmacokinetics and pharmacodynamic profile of CBD in normal healthy individuals under standard and high fat fed conditions.

CBD has recently gained significant attention as a potential treatment for various disorders. One aspect for consideration in the development of CBD medication in capsule form is the poor bioavailability of cannabinoids such as CBD to obtain clinically effective doses since only ~4-6% of CBD is absorbed orally. This study will investigate the potential of CBD in a formulation in a capsule to enhance bioavailability, reduce the incidence of gastrointestinal side effects, reduce first pass metabolism and enhance onset time. This PK study will be conducted with standard meal and high fat conditions in normal healthy volunteers in a cross-over design, separated by a washout period of 1 week. Healthy volunteers are defined as having no significant health-related issues (i.e., the absence of significant medical, psychosocial, or emotional conditions) that are verified by clinical and psychiatric assessments.

The study will first evaluate in healthy volunteers the PK, tolerability and safety profiles of a new CBD formulation designed to improve bioavailability.

Test conditions and order:

1. 200 mg CBD (standard meal)
2. 400 mg CBD (standard meal)
3. 400 mg Epidiolex (standard meal)
4. 400 mg CBD (high fat meal)

Blood samples will be taken at -60,15, 30, 45 and 60 min and1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours associated with administration of the CBD capsules.

Monitoring period for PK: 24 hours (plasma and urine PK). Participation in 4 test conditions for a duration of approximately 4 weeks and a 1-week follow-up assessment.

Total length of in-house stay is 12 hours, with participants returning the following day for 24-hour time point procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent;
* Individuals between 18 and 65 years old; Sex is used a biological factor (50% of individuals recruited will be females, allowing sex comparisons).
* English speakers.
* Being healthy as determined by study physician according to screening medical and psychiatric history, physical examination, vitals, ECG and safety laboratory values. Only healthy volunteers with normal hepatic laboratory values will be enrolled.
* Healthy volunteers who are medication- and drug-free, including free from nicotine and any prescribed medications.

Exclusion Criteria:

* Having present or past medical conditions, including a DSM-5 Axis I psychiatric disorder, history of cardiac disease, arrhythmias, neurological disease of central origin, head trauma, and seizures
* Using any psychoactive drug (other than nicotine) in at least the past 7 days (determined by lack of acute-opioid or other drugs related withdrawal symptoms and the negative result of a urine drug screen including an opioid drug metabolite test, and alcohol breathalyzer to detect alcohol intoxication);
* Positive urine drug screen (cocaine, opiates, benzodiazepines, barbiturates, amphetamines, morphine, methadone, methamphetamines, oxycodone, phencyclidine, tricyclic antidepressant, tetrahydrocannabinol, buprenorphine, methylenedioxymethamphetamine, propoxyphene);
* Having a history of hypersensitivity to cannabinoids or any of the ingredients in the product (gelatin and/or sesame oil);
* Being pregnant or breastfeeding;
* Not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e. condom, spermicide, diaphragm);
* Participating in another pharmacotherapeutic trial in the past 3 months;
* History of impaired renal function or elevated liver enzymes at prescreening. The exclusionary lab values are: 3x nl AST/ALT, 1.5x bilirubin or 50%reduction in eGFR.
* Participants who have used any medication, dietary supplements (and/or grape fruit juice), or combination of medications and supplements known to alter the metabolism of, or interact with CBD (bupropion, rifampin, barbiturates, phenothiazines, cimetidine, etc.) 14 days prior to and during the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Systematic Assessment for Treatment Emergent Events (SAFTEE) | up to 24 hours post-treatment
  Systematic Assessment for Treatment Emergent Events (SAFTEE) to measure safety and adverse events.
Peak Plasma Concentration (Cmax) | up to 24 hours post-treatment
  Peak plasma concentration of CBD and its metabolites
Area under the plasma concentration curve (AUC) | up to 24 hours post-treatment
  Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
Peak urine concentration of CBD (Umax) | up to 24 hours post-treatment
  Peak urinary excretion of CBD and its metabolites
Area under the urine concentration curve (AUC) | up to 24 hours post-treatment
  Area under the urine concentration versus time curve

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States